CLINICAL TRIAL: NCT04855409
Title: Neuronal Integrity and Suicidality in Bipolar Depression: a Diffusion Tensor Imaging Study
Brief Title: Neuronal Integrity in Bipolar Depression
Status: Completed | Type: Observational
Sponsor: Mehmet Diyaddin Güleken (Other)
Responsible Party: Sponsor-Investigator, Mehmet Diyaddin Güleken, Attending Physician, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: 21012021
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Bipolar I Disorder, Most Recent Episode Depressed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar Depression: Subjects with bipolar type I disorder depressive episode diagnosed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I)
- Healthy: Healthy control subjects matched with bipolar depressive patients by age and sex

SUMMARY:
The aim of this study is to examine the neurological unity in bipolar depression and to investigate white matter abnormalities that may contribute to etiology

DETAILED DESCRIPTION:
Bipolar disorder is a chronic mood disorder which is characterized by repetitive episodes, usually manifests through adolescence or early adulthood. It has a prevalence of approximately 2,5% with a 1:1 ratio of male and female. It is a disorder that may disrupt central nervous system functions such as cognition, thought, perception, affect, judgement, adaptation to the environment and behavioural regulation. It may manifest with various clinical onsets. Although etiology of bipolar disorder is still unknown, some biological factors such as BDNF, oxidative stress and structural changes of brain are proven to have a role in etiology.

Diffusion tensor magnetic resonance imaging (DTI) is a neuroimaging technique that elucidates abnormalities of brain white matter (WM), based on structural investigation of a tissue via measurement of diffusion rate and direction of water molecules. This method lets imaging of white matter tracts, whole anatomical extent and structural integrity of the brain tissue. So, it can provide data about anatomical connectivity of brain. There are some parameters used for indicating microstructural integrity of white mat-ter such as fractional anisotropy (FA) and apparent diffusion coefficient (ADC) in DTI. FA is a measure which reflects directional coherence of water diffusion, and it is sen¬sitive to microstructural WM differences. It is defined on a scale ranging from mostly isotro¬pic (when approaching to zero) indicating poor integrity of the axons to mostly anisotropic (when approaching to 1) indicating intact WM integrity. ADC is a scalar index of the rate of water diffusion among different dif¬fusion directions under a Gaussian distribution. A higher value of ADC indicates lesser restricted diffusion, and it implies fewer organized structures in WM which supports presence of abnormalities in the structural in¬tegrity of white matter. As it has a complicated literature, in this study, we aimed to investigate neuronal integrity and its abnormalities by DTI, which may contribute to the etiology of bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* Aged between 18 and 65
* Having a diagnosis of bipolar type I disorder depressive episode by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I)
* Having no other general medical, neurological or psychiatric condition Healthy controls;
* Matched with bipolar depressive patients by age and sex
* Having no other general medical, neurological and psychiatric condition

Exclusion Criteria:

* Bipolar depressive patients and healthy control subjects with any other general medical, neurological or psychiatric condition, metal implant, severe head injury or pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sixteen subjects with bipolar type I disorder depressive episode diagnosed by SCID-I were recruited from Psychiatry Department of Harran University Research Hospital, and sixteen healthy control subjects were enrolled from the hospital staff. Patient and control groups have been matched by age and sex. A written informed consent was obtained from each volunteered participant.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Brain white matter abnormality | Within a day
  The fractional anisotropy and appearent diffusion coefficient parameters of corpus callosum genu and corpus callosum splenium of both groups

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Çelik, MD, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan about sharing individual participant data with other researchers